CLINICAL TRIAL: NCT01693835
Title: Molecularly Imprinted Polymer Sensors of Modified Nucleosides for Non-invasive Monitoring of Cancer Therapy : the Circadian Rhythms of Urinary Excretion of Modified Nucleosides.
Brief Title: "Cancersensor": Circadian Rhythms
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C11-42; 2012-A00010-43 (Registry Identifier: IDRCB)
Record Dates: First submitted 2012-09-07; First posted 2012-09-26 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2016-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal; Cancer; Metastatic; Healthy; Control; Circadian; Urine; Nucleosides
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva (exfoliated oral mucosa cells) and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: Patients with metastatic colorectal cancer
- Healthy subjects: Age and sec-matched healthy subjects

SUMMARY:
Observational, non randomized study aimed at measuring the circadian rhythms in the urinary concentrations of physiological modified nucleosides in 30 patients with metastatic colorectal cancer and in 30 age and sex-matched healthy subjects.

ELIGIBILITY:
Inclusion Criteria for patients:

* Histologically-confirmed metastatic colorectal cancer;
* 0 to 3 prior chemotherapy lines;
* Signed informed consent;
* Good understanding of the protocol and of the follow-up;
* Estimated life expectancy exceeding 3 months;
* At least one measurable metastatic lesion (RECIST criteria);
* Performance Status (WHO) of 0 to 2;
* Good haematological, hepatic and renal functions.

Inclusion criteria for healthy subject

* Age ≥ 18 ans
* Signed informed consent;
* Good understanding of the protocol and of the follow-up;
* Good haematological, hepatic and renal functions.
* Test HIV and B and C hepatitis negative test
* No chronic or acute diseases

Exclusion Criteria for patients:

* Poor performance status (>2);
* Poor haematological, hepatic or renal functions;
* Uncontrolled chronic disease;
* Serious unhealed wound, ulcer or fracture within the previous month;
* Clinical or laboratory finding suggesting possible abnormalities in nucleosides urinary excretion;
* Pregnancy or breast-feeding during the previous month;
* Transmeridian trip of more than 4 time zones within the prior 2 weeks;
* Person with legal restriction to participate into clinical research, according to the current law in France.

Exclusion criteria for healthy subject:

* Poor haematological, hepatic or renal functions;
* Uncontrolled chronic disease;
* Serious unhealed wound, ulcer or fracture within the previous month;
* Clinical or laboratory finding suggesting possible abnormalities in nucleosides urinary excretion;
* Pregnancy or breast-feeding during the previous month;
* Transmeridian trip of more than 4 time zones within the prior 2 weeks;
* Person with legal restriction to participate into clinical research, according to the current law in France.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic colorectal cancer treated at the Department of Medical Oncology of Paul Brousse Hospital
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Circadian rhythms in urinary excretion of modified nucleosides | 2 days repeated measures
  10 Urine samples over 2 days Measurement of modified nucleosides, cortisol and 6-sulfatoxymelatonin concentration
  1 saliva sample Measurement of Clock genes polymorphisms expression

CONTACTS AND LOCATIONS:
Overall Officials: Francis Lévi, MD, PhD, Principal Investigator — INSERM and AP-HP and Paris South University; Sandrine Dulong, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Paul Brousse Hospital, Villejuif, France

REFERENCES:
- [Result] Dulong S, Huang Q, Innominato PF, Karaboue A, Bouchahda M, Pruvost A, Theodoro F, Agrofoglio LA, Adam R, Finkenstadt B, Levi F. Circadian and chemotherapy-related changes in urinary modified nucleosides excretion in patients with metastatic colorectal cancer. Sci Rep. 2021 Dec 14;11(1):24015. doi: 10.1038/s41598-021-03247-2. PMID 34907230